CLINICAL TRIAL: NCT05993494
Title: Investigation of the Relationship Between Pain, Central Sensitization, Kinesiophobia and Stress Level in Individuals With Temporomandibular Dysfunction
Brief Title: Pain, Central Sensitization, Kinesiophobia and Stress Level in Individuals With Temporomandibular Dysfunction
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Research assistant, Karadeniz Technical University
Other Study IDs: KTU-FTR-2023/6
Record Dates: First submitted 2023-07-30; First posted 2023-08-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Joint Disorders; Pain
Keywords: Temporomandibular Joint Dysfunction; Pain; central sensitization; kinesiophobia; stress
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Temporomandibular dysfunction (TMD) is a musculoskeletal and neuromuscular system-related condition that affects the masticatory muscles, temporomandibular joint, and other related structures. Recent research has focused specifically on pain catastrophe, kinesiophobia, and central sensitization in individuals with TMD. Therefore, the aim of this study is to examine the relationship between pain, central sensitization, kinesiophobia and stress level in individuals with temporomandibular dysfunction.

DETAILED DESCRIPTION:
Temporomandibular dysfunction (TMD) is a musculoskeletal and neuromuscular system-related condition that affects the masticatory muscles, temporomandibular joint, and other related structures. Psychological factors are stated as comorbid in individuals with TMD. Individuals with TMD-related pain show higher levels of stress, anxiety, depression, somatic awareness, pain catastrophizing, and kinesiophobia compared to controls. Therefore, recent research has focused on pain catastrophe, kinesiophobia, and central sensitization, especially in individuals with TMD. Therefore, the aim of this study is to examine the relationship between pain, central sensitization, kinesiophobia and stress level in individuals with temporomandibular dysfunction. Ninety patients aged 18-65 years, who have TME-related complaints for at least 3 months, and diagnosed with TMD as a result of clinical and radiological evaluation by a dentist will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Having complaints related to TMJ for at least 3 months,
* Patients diagnosed with TMD as a result of clinical and radiological evaluation by the dentist

Exclusion Criteria:

* Cognitive problems,
* Any systemic joint or muscle disease (e.g. fibromyalgia, rheumatoid arthritis),
* Serious systemic diseases,
* Any neurological disorder (e.g. trigeminal neuralgia),
* Pregnancy, breastfeeding status,
* Previous treatment for TMJ or orofacial muscle pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Patients diagnosed with Temporomandibular joint disorders
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Scale | through study completion, an average of 1 year
  Pain Assessment
Tampa Scale for Kinesiophobia | through study completion, an average of 1 year
  Kinesiophobia Assessment for temporomandibular joint dysfunction
Perceived Stress Scale | through study completion, an average of 1 year
  Stress Assessment
Central sensitization scale | through study completion, an average of 1 year
  Central sensitization Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nurhayat Korkmaz, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No